CLINICAL TRIAL: NCT00000729
Title: A Multicenter Study To Determine Foscarnet Dose Response in HIV Infected Patients With PGL and/or Constitutional Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: ACTG 028; 11004 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Virus Replication; Infusions, Intravenous; Dose-Response Relationship, Drug; Foscarnet; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; CD4-Positive T-Lymphocytes
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Foscarnet

INTERVENTIONS:
Drug: Foscarnet sodium

SUMMARY:
To determine the toxicity of low dose foscarnet administered for 4 weeks to HIV infected patients who are asymptomatic, have AIDS, or other HIV associated conditions and a CD4+ lymphocyte count < 500 cells/mm3. To obtain preliminary efficacy data. Although zidovudine (AZT) has been effective in treating some AIDS patients, AZT has toxic effects in many patients and other means of treating HIV-infected persons need to be evaluated. In vitro (test tube) studies have shown that the human herpes viruses are inhibited by foscarnet and that a number of retroviruses, including HIV, are sensitive to it. It is hoped that treatment of HIV-infected individuals with foscarnet during an early phase of HIV infections will reduce the risk of developing AIDS.

DETAILED DESCRIPTION:
Although zidovudine (AZT) has been effective in treating some AIDS patients, AZT has toxic effects in many patients and other means of treating HIV-infected persons need to be evaluated. In vitro (test tube) studies have shown that the human herpes viruses are inhibited by foscarnet and that a number of retroviruses, including HIV, are sensitive to it. It is hoped that treatment of HIV-infected individuals with foscarnet during an early phase of HIV infections will reduce the risk of developing AIDS.

Patients are divided into three groups: (1) asymptomatic patients with or without persistent generalized lymphadenopathy (PGL) syndrome; (2) patients with AIDS; and (3) patients who have or have had mild to moderate signs or symptoms consistent with HIV infection. Patients are then randomly chosen to receive one of three different foscarnet doses. The drug is given for 4 weeks, by 1-hour infusion administered every 8 hours. In addition, those patients who are clinically stable and have not experienced severe toxicity at the end of the 4 weeks may continue treatment, in the form of a single daily dose of foscarnet to be administered 5 days per week. Blood samples are taken during treatment and at the first, fourth, and eighth week after treatment. If the patient is on maintenance, blood samples are taken weekly. Effective 7-17-89, patients entering the study are assigned to the lowest foscarnet dose. Patients receive daily treatment for 28 days. Patients who are clinically stable without severe toxicity at 4 weeks have the option of maintenance therapy with foscarnet.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Aerosolized pentamidine for secondary Pneumocystis carinii pneumonia (PCP) prophylaxis.
* Short course therapy with oral acyclovir (ACV) = or < 7 days. Short course therapy with ketoconazole = or < 7 days for patients who are not responding to any other therapy.
* Flurazepam.
* Diphenhydramine.

Prior Medication:

Allowed:

* Systemic therapy, prophylaxis or maintenance for an AIDS-defining opportunistic infection.

Patients with any of the following findings may be included:

* Asymptomatic HIV patients with or without lymphadenopathy.
* Patients with AIDS as defined by the CDC surveillance case definitions.
* Patients with past or present mild to moderate signs or symptoms consistent with HIV infection.
* p24 antigen in the serum = or > 60 pg/ml.

Exclusion Criteria

Co-existing Condition:

Patients with the following will be excluded:

* Ongoing systemic therapy / prophylaxis / maintenance for an AIDS-defining opportunistic infection.
* Symptomatic visceral Kaposi's sarcoma (KS), progression of KS within the month prior to entry into the study, or with concurrent neoplasms other than KS or basal cell carcinoma of the skin or in situ carcinoma of the cervix.
* Cytomegalovirus (CMV) retinitis.
* AIDS dementia.

Concurrent Medication:

Excluded:

* Antiretrovirals.
* Immunomodulatory agents.
* Corticosteroids Other systemic antiviral or antimicrobial agents.
* Experimental medications.
* Excluded on chronic basis and discouraged for > 72 hours:
* Acetaminophen.
* Narcotics.
* Aspirin.

Concurrent Treatment:

Excluded:

* Transfusion dependency or requirement of 2 units of blood more than once per month.

Patients with the following will be excluded:

* Ongoing systemic therapy / prophylaxis / maintenance for an AIDS-defining opportunistic infection.
* Symptomatic visceral Kaposi's sarcoma (KS), progression of KS within the month prior to entry into the study, or with concurrent neoplasms other than KS or basal cell carcinoma of the skin or in situ carcinoma of the cervix.
* Cytomegalovirus (CMV) retinitis.
* AIDS dementia.

Prior Medication:

Excluded within 30 days of study entry:

* Antiretroviral agents (except ribavirin).
* Immunomodulatory agents.
* Excluded within 60 days of study entry:
* Ribavirin.

The last blood transfusion cannot have been given within 2 weeks of entry.

Active substance abuse which could impair compliance with the protocol.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10
Dates: Study Completion 1992-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Collier AC, Study Chair
Locations (11):
- United States (11):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - USC School of Medicine / Norris Cancer Hosp, Los Angeles, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Univ of Minnesota, Minneapolis, Minnesota
  - City Hosp Ctr at Elmhurst / Mount Sinai Hosp, Elmhurst, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - SUNY - Stony Brook, Stony Brook, New York
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Background] Fletcher CV, Collier AC, Rhame FS, Bennett D, Para MF, Beatty CC, Jones CE, Balfour HH Jr. Foscarnet for suppression of human immunodeficiency virus replication. Antimicrob Agents Chemother. 1994 Mar;38(3):604-7. doi: 10.1128/AAC.38.3.604. PMID 7911290